CLINICAL TRIAL: NCT02940444
Title: Safety and Efficacy of Preoperative Administration of Heparin as Thromboprophylaxis in Major Thoracic Surgery
Brief Title: Preoperative Administration of Heparin as Thromboprophylaxis in Major Thoracic Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yi-Dan Lin, proffessor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WCH-20160601
Record Dates: First submitted 2016-10-17; First posted 2016-10-21 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Thromboprophylaxis; Thoracic Surgery
MeSH Terms: interventions — Heparin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- case group (Experimental): start heparin sodium (5000IU, BID) upon admission, and continue until discharge
  Interventions: Drug: Heparin
- control group (Active Comparator): start heparin sodium (5000 IU,BID) from postoperative day 1, and continue until discharge
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Heparin

SUMMARY:
Thromboembolism is an important perioperative complication in major thoracic surgery, even though current guidelines have recommended postoperative administration of heparin or LMWH for thromboprophylaxis for those high-risk patients, there are still many cases of thromboembolism. Therefore, as the guideline itself writes, the investigators believe the rational of dose and timing of heparin in thoracic surgery are still not well established. Therefore, the investigators aimed to conduct this randomized controlled study to explore the safety and efficacy of preoperative Administration of Heparin as Thromboprophylaxis in Major Thoracic Surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old without any preoperative VTEs;
* patients undergoing major thoracic surgery (including lobectomy, esophagectomy, and thymectomy).

Exclusion Criteria:

* patients with coagulation disorders: preoperative international normalized ratio (INR) > 1.5, or blood platelet count < 50x10^9/L;
* patients receiving any therapeutic anticoagulation preoperatively;
* patients with severe renal or liver dysfunction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
intraoperative bleeding volume (ml) | the bleeding volume (ml) during operation in the operation room for all patients
  During the operation, the blood loss of each patient was collected and measured, and recorded by the investigators.
chest tube drainage volume (ml) | from postoperative day 1 to chest tube remove(usually on postoperative day 3 for lobectomy or thymectomy,on postoperative day 7 for esophagectomy )
thromboembolism occurence rate (%) | within 30 days after surgery
APTT (s) | on postoperative day 1 for both group
PT(s) | on postoperative day 1 for both group
INR | on postoperative day 1 for both group
blood platlet count(/L) | on postoperative day 1 for both group
chest tube drainage duration (days) | from postoperative day 1 to chest tube remove(usually on postoperative day 3 for lobectomy or thymectomy,on postoperative day 7 for esophagectomy )

SECONDARY OUTCOMES:
PT(s) | rightly upon hospital admission day
APTT(s) | rightly upon hospital admission day
INR | rightly upon hospital admission day
blood platlet count(/L) | rightly upon hospital admission day

CONTACTS AND LOCATIONS:
Locations (1):
- Department of thoracic surgery, west china hospital, sichuan university, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Deng HY, Shi CL, Li G, Luo J, Wang ZQ, Lin YD, Liu LX, Zhou QH. The safety profile of preoperative administration of heparin for thromboprophylaxis in Chinese patients intended for thoracoscopic major thoracic surgery: a pilot randomized controlled study. J Thorac Dis. 2017 Apr;9(4):1065-1072. doi: 10.21037/jtd.2017.03.148. PMID 28523161